CLINICAL TRIAL: NCT04208932
Title: A Kynurenine Pathway-based Molecular Imaging Study of Individualized Diagnosis and Treatment for Major Depressive Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: ZH2018ZDA29
Record Dates: First submitted 2019-12-20; First posted 2019-12-23 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MDD: major depressive disorder
  Interventions: Drug: SSRIs
- HC: healthy control

INTERVENTIONS:
Drug: SSRIs — Selective Serotonin Reuptake Inhibitors
  Groups: MDD

SUMMARY:
Major depressive disorder (MDD) is a chronic disease with high incidence rate, high recurrent rate and need whole course medical management. Varied clinical symptoms and unclear pathogenesis cause a series of clinical problem, such as low diagnostic rate and low effective treatment rate. Based on neuroimmune mechanisms of MDD, our previous study indicates that kynurenine pathway (KP) in serum may be the connections between central immune and peripheral immune, that key factors of KP may change the brain structure and function through affecting the central immune. The core research issue of this project are the inherent associations between metabonomics of inflammatory factors in KP, clinical phenotypes of MDD, and neuroimaging features. This project will focus on first-episode MDD, mass spectrometry analysis of KP factors will be conducted first, also multi-modal neuroimaging techniques will be applied to detect topological characteristics of brain structure and function in MDD and extract standard models, then correlation analyses will be performed between these molecular biological features and multi-dimensional clinical data in order to integrate KP metabonomics, core clinical characteristics (depressed mood, energy loss, interest loss and so on), neuroimaging biomarkers, and finally construct the deep learning based standard diagnostic technique of MDD. Additionally, this project will follow up MDD patients with different core clinical characteristics to certificate the aforementioned diagnostic technique as well as explore optimized treatment for different clinical subtypes.

ELIGIBILITY:
Inclusion Criteria:

1. 18-60 years old;
2. Meeting with the criteria of major depressive disorder in the Diagnostic and Statistical Manual of Mental Disorders (DSM)-5;
3. Scored 20 or higher on the Hamilton's Depression Scale with 24 items (HAMD-24);
4. With enough audio-visual ability and comprehensive ability to accomplish the visits;
5. Be necessary and suitable to accept the treatment of antidepressants;
6. Scored less than 14 on Hamilton's Anxiety Scale (HAMA) and scored less than 14 on the Hypomania Symptom Checklist-32 (HCL-32);
7. With 2 or more atypical symptoms including significant weight gain or increase in appetite, hypersomnia, leaden paralysis, and a long-standing pattern of interpersonal rejection sensitivity that results in significant social or occupational impairment.

Exclusion Criteria:

1. Severe medical or neurological problems;
2. Previous mania or hypomania episodes;
3. Female patients who are pregnant, planning to be pregnant or breastfeeding;
4. Actively suicide ascertained by research psychiatrist or 3rd item of HAMD scored≥3(suicidality);
5. Had electroconvulsive therapy, modified electroconvulsive therapy or repetitive transcranial magnetic stimulation in the past 6 months;
6. Experienced severe personality disorder, mental retardation, anorexia/bulimia nervosa.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 370 patients with the major depressive disorder who are first-episode drug-naive or medication-free for no less than 2 weeks; 70 healthy participants
Sampling Method: Non-Probability Sample
Enrollment: 440 (Estimated)
Dates: Start 2019-08-12 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
remission of acute phase | 12th week
  scored 7 or lower on the Hamilton's Depression Scale with 24 items

CONTACTS AND LOCATIONS:
Overall Officials: Daihui Peng, MD.PhD., Study Chair — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided